CLINICAL TRIAL: NCT04124718
Title: Association Between Enamel Gene Variants and Dental Caries in Adults
Brief Title: VDR and TFIP11 Gene Polymorphism and Gene-environmental Interaction in Adults
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2019-204
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Low Caries Experience; High Caries Experience
Keywords: caries experience, VDR, TFIP11, enviromental risk factor
MeSH Terms: interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — DNA for genetic analysis was isolated from buccal epithelial cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high caries experience: 80 adults will be allowed in the high caries experience group according to DMFT index DMFT>13.9
  Interventions: Genetic: high caries experience
- low caries experience: 80 adults will be allowed in the high caries experience group according toDMFT index DMFT≤4
  Interventions: Genetic: high caries experience

INTERVENTIONS:
Genetic: high caries experience — DNAs were obtained from epithelial cells in buccal mucosa and were extracted with Genomic DNA Isolation Kit
  Other Names: DNA isolation, genotyping

SUMMARY:
VDR and TFIP11 Gene polymorphism and gene-environment interactions on caries etiology and susceptibility in adults.

DETAILED DESCRIPTION:
To date, genes can be grouped into categories based on the factor influencing dental caries. The major candidate gene categories to date include enamel formation genes, immune response genes, genes related to saliva, and genes related to taste and dietary habits.

TFIP11 and VDR genes are related to enamel formation genes

ELIGIBILITY:
Inclusion Criteria:

* adult be between 24 and 40 years old
* subject has DMFT (Decayed, Missing, Filled, Permanent Tooth) DMFT≤4 , or, DMFT>13.9

Exclusion Criteria:

* systemic or genetic disorders
* orthodontic appliances
* pregnant women

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 160 adult in the 24-40 age range living in Northeast Turkey will allowed in the study
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
past caries experience | 3 weeks
  Each tooth will be examined and recorded as decayed, missing, or filled

SECONDARY OUTCOMES:
Plaque index | 3 weeks
  The plaque amount is scored by using Silness&Löe Plaque Index plaque index PI<1.0 healthy PI 1.1-2.0 mild PI>2 high plaque

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yıldız Telatar, dr, Principal Investigator — Recep Tayyip Erdogan University Dentistry Faculty
Locations (1):
- Recep Tayyip Erdogan University Dentistry Faculty, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be available within 6 months of study completion

REFERENCES:
- [Background] Cogulu D, Onay H, Ozdemir Y, Aslan GI, Ozkinay F, Eronat C. The Role of Vitamin D Receptor Polymorphisms on Dental Caries. J Clin Pediatr Dent. 2016;40(3):211-4. doi: 10.17796/1053-4628-40.3.211. PMID 27472568
- See also: The Role of Vitamin D Receptor Polymorphisms on Dental Caries. — http://www.ncbi.nlm.nih.gov/pubmed/27472568